CLINICAL TRIAL: NCT06611267
Title: En undersøgelse af Smerteoplevelsen Hos Raske forsøgsdeltagere (A Study of the Pain Experience in Healthy Participants)
Brief Title: Experiences of Pain in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: EXPERIENCES OF PAIN
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Pain in Healthy Adults
Keywords: Healthy adults; Pain; Experience of pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants assess their experienced pain (Experimental)
  Interventions: Other: Pain without cream on; Other: Pain with cream on
- Participants assess their expected and experienced pain (Active Comparator)
  Interventions: Other: Pain without cream on; Other: Pain with cream on

INTERVENTIONS:
Other: Pain without cream on — Participants will be inflicted with pain without cream on.
Other: Pain with cream on — Patients are inflicted with pain after getting a cream on, which has previously had pain-relieving effects

SUMMARY:
The experiment aims to investigate the experience of pain in healthy adults and includes a total of 60 participants. Pain is a subjective experience that has a complicated neurological and psychological basis. Around 20% of the Danish population suffers from persistent pain, which has both personal and societal consequences. Personal consequences include, among others, reduced quality of life, loss of social life and risk of anxiety and depression. However, more knowledge is needed about which mechanisms are involved in the experience of pain, so that the treatment of patients with pain can be improved.

In the experiment, healthy participants will be inflicted with a tolerable pain on their forearm using a thermode. The application of heat causes pain for a short, limited period, but it is tolerable and without risks. During the experiment, the participants will be exposed to heat several times, with and without a cream on their forearm. It is a cream that has previously proved to have pain-relieving effects on participants in similar experiments. Participants will be asked about how they experience the intensity of the pain on a scale of 1-10 (0 = no pain and 10 = worst imaginable pain), and what they expect the pain intensity will be, also on a 1-10 scale. The participants are allowed to pause or stop the experiment anytime.

The experiment contributes to insights into pain and the mechanisms involved. This knowledge can in the future contribute with knowledge to improve the treatment of patients with pain. For the individual participant, the trial will contribute with knowledge about how they experience and assess pain themselves.

ELIGIBILITY:
Inclusion Criteria:

* Normal health, i.e. no known acute or chronic illness
* Fluid in Danish

Exclusion Criteria:

* Chronic pain condition
* Other medical or psychiatric disorder
* Use of antidepressants
* Daily use of painkillers
* Use of pain medication 24 hours prior to testing
* Drug abuse
* Pregnancy
* Studying or with completed education in psychology or journalism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2025-02-07 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Experienced pain measured on a Visual Analogue Scale (VAS) from 0-10 (from no pain to worst imaginable pain) without cream compared to experienced pain measured on a Visual Analogue Scale (VAS) from 0-10 (from no pain to worst imaginable pain) with cream | From beginning to end of experiment, approx. 45 minutes

SECONDARY OUTCOMES:
The effect of assessing expected pain intensity measured on a Visual Analogue Scale (VAS) from 0-10 (from no expected pain to worst imaginable expected pain) | From beginning to end of experiment, approx. 45 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No